CLINICAL TRIAL: NCT07077772
Title: Evaluation of Natriuresis-guided Depletion After Cardiac Surgery: a Monocentric, Open-label, Randomized Controlled Trial
Brief Title: Natriuresis-guided Depletion After Cardiac Surgery
Acronym: EASY-CS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Principal Investigator, Beyls, Principal Investigator, Centre Hospitalier Universitaire, Amiens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2025_843_0080
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery; Diuresis; Congestion, Venous; Sodium Depletion; Fluid Over-load
Keywords: natriuresis; fluid overload; cardiac surgery; furosemide; venous congestion; loop diuretics
MeSH Terms: conditions — Hyperemia; Hyponatremia; Edema

STUDY DESIGN:
Intervention Model Description: Furosemide IV, 20 mg starting dose, titrated every 6 hours based on urinary sodium (experimental) or clinical evaluation (control)
  The investigators predefined safety criteria to be assessed prior to each furosemide injection in order to monitor potential complications related to its administration, including:
  * Symptomatic hypotension, defined as a mean arterial pressure < 65 mmHg requiring fluid resuscitation or vasopressor support;
  * Hypokalemia, defined as a serum potassium concentration < 3 mmol/L;
  * Impaired renal function, defined as a doubling of serum creatinine or a ≥50% decrease in estimated glomerular filtration rate (eGFR) within the first 48 hours.
  The study protocol will be implemented over a 48-hour timeframe starting from patient inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natriuresis-Guided Arm (Experimental): Furosemide IV, 20 mg starting dose, titrated every 6 hours based on urinary sodium measured by the LAQUATWIN device.
  Interventions: Drug: Furosemide intravenous titration based on natriuresis
- Control (Active Comparator): Furosemide IV, 20 mg starting dose, titrated every 6 hours based on clinical evaluation
  Interventions: Drug: Furosemide intravenous titration based on clinical examination

INTERVENTIONS:
Drug: Furosemide intravenous titration based on natriuresis — Furosemide IV, 20 mg starting dose, titrated every 6 hours based on urinary sodium measured by the LAQUAtwin NA-11 device.
  Urine output will be measured and recorded every 4 hours to ensure accurate diuresis tracking.
  If natriuresis is < 70 mmol/L, the furosemide dose will be doubled, with a maximum limit of 200 mg per bolus.
  If natriuresis is ≥ 70 mmol/L, the current dose will be maintained.
  Blood electrolyte panels and renal function assessments will be performed twice daily throughout the protocol.
  In the event of hemodynamic instability, a complete echocardiographic assessment will be performed for all patients to detect potential surgical complications, along with a hemodynamic evaluation to guide appropriate management.
  Arms: Natriuresis-Guided Arm
Drug: Furosemide intravenous titration based on clinical examination — Furosemide IV, 20 mg starting dose, titrated every 6 hours clinical evaluation.
  Urine output will be measured and recorded every 4 hours to ensure accurate diuresis tracking.
  The furosemide dosage will be adjusted based on urine output with a maximum bolus dose of 200 mg. Dose adjustments will be reassessed every 6 hours throughout the study period.
  Blood electrolyte panels and renal function assessments will be performed twice daily throughout the protocol.
  In the event of hemodynamic instability, a complete echocardiographic assessment will be performed for all patients to detect potential surgical complications, along with a hemodynamic evaluation to guide appropriate management.
  Arms: Control

SUMMARY:
Fluid overload (FO) is a common complication after cardiac surgery, associated with increased morbidity and mortality. Loop diuretics, especially furosemide, are routinely used to manage FO, but their use is often empirical. Recent data suggest that natriuresis-guided furosemide titration using point-of-care urinary sodium sensors (LAQUAtwin NA-11, Horiba) may improve the efficiency and safety of fluid removal, but no randomized trial has yet evaluated this approach in postoperative cardiac surgery patients

Our goal is to assess the clinical impact, safety, and feasibility of a natriuresis-guided furosemide protocol after cardiac surgery requiring cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age > 18 years)
* Scheduled for cardiac surgery, including mitral valve repair or replacement, aortic valve replacement, coronary artery bypass grafting (CABG), ascending aortic repair, or combined procedures
* Undergoing surgery with cardiopulmonary bypass (CPB)
* Eligible to receive intravenous furosemide for fluid overload within 48 hours following surgery, as prescribed by the referring physician
* Written and oral informed consent obtained
* Covered by the French national health insurance (Sécurité Sociale)

Exclusion Criteria:

* Aortic arch repair requiring deep hypothermic circulatory arrest
* Active endocarditis
* Hemodynamic instability requiring vasopressor or inotropic support (norepinephrine, dobutamine, epinephrine, or vasopressin)
* Failure to wean from CPB requiring mechanical circulatory support
* Chronic kidney disease with an estimated glomerular filtration rate (eGFR) < 60 mL/min
* Chronic use of loop diuretics
* Known allergy to furosemide
* Active postoperative bleeding and/or reoperation for bleeding
* Participation in another interventional study that may affect the primary outcome measure
* Patient deprived of liberty by administrative or judicial decision, or placed under legal protection (guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Total urine output (mL) at 48 hours after randomization. | 48 hours after randomization
  All patients were equipped with urinary catheters, allowing for continuous urine collection. Urine output was measured every 2 hours, and the recorded volumes were entered into a monitoring software to ensure accurate follow-up

SECONDARY OUTCOMES:
Urine output at 24 hours | 24 hours after randomization
  All patients were equipped with urinary catheters, allowing for continuous urine collection. Urine output was measured every 2 hours, and the recorded volumes were entered into a monitoring software to ensure accurate follow-up.
Natriuresis at 24 hours | 24 hours after randomization
  Total natriuresis is measured at 24 hours using the indirect potentiometry technique at the CHU Amiens-Picardie laboratory.
Natriuresis at 48 hours | 48 hours after randomization
  Total natriuresis is measured at 48 hours using the indirect potentiometry technique at the CHU Amiens-Picardie laboratory.
VExUS score at 48 hours | 48 hours after randomization
  The VExUS score is an echocardiographic score (ranging from 0 to 3) used to assess venous congestion at the cardiac, renal, and hepatic levels. This score will be measured after randomization and at 48 hours after randomization.
  Grade 0: IVC <2cm = No Congestion Grade 1: IVC >2cm with any combo of Normal or Mildly Abnormal Patterns = Mild Congestion Grade 2: IVC >2cm and one severely Abnormal Pattern = Moderate Congestion Grade 3: IVC >2cm and >2 Severely Abnormal Patterns = Severe Congestion
Total loop diuretics | During the study period (48 hours)
  Total dose of loop diuretics administered during the study period (mg)
Cumulative Fluid balance | At inclusion and 48 hours after randomization
  Fluid balance corresponds to the difference between administered fluids (intravenous infusions, blood products, enteral nutrition) and fluid losses (urine output, blood loss, digestive losses, drain output). It is calculated using the DianeRéa software (Bowmedical, version 4.8.11.22887), taking into account all fluid inputs (administered fluids, medications, nutrition) and all fluid outputs (urine, drains, perspiration) over the period from inclusion to 48 hours after randomization
Number of Participants with Postoperative Complications by Day 30 | Day 30 after randomization
  Composite outcome measuring the number of participants who experience at least one of the following postoperative complications within 30 days of surgery:
  Cardiovascular:
  * Acute left and right ventricular systolic heart failure
  * Acute circulatory failure requiring catecholamine support
  * Supraventricular (e.g., atrial fibrillation) or ventricular arrhythmias.
  Respiratory:
  * Acute respiratory distress syndrome (ARDS)
  * Prolonged orotracheal intubation (> 24 hours).
  * Reintubation.
  Renal:
  - Acute kidney injury (AKI), defined by a postoperative increase in serum creatinine of at least 50% and/or ≥ 26.5 µmol/L from baseline, and/or urine output < 0.5 mL/kg/h for ≥ 6 hours (KDIGO criteria). Serum creatinine and estimated glomerular filtration rate (eGFR) measured on the day of hospital discharge.
  Gastrointestinal:
  * Mesenteric ischemia or ischemic colitis, documented by imaging (CT scan), colonoscopy, and/or surgery.
  * Length of hospital stay (days).
  * In-hospital mortality.
Number of Participants with Contraindications to Furosemide Administration | During the study period (48 hours after randomization)
  Number of participants presenting contraindications prior to furosemide administration, including:
  * Symptomatic hypotension
  * Hypokalemia
  * Impaired renal function
Number of Corrective Measures Implemented Prior to Furosemide Administration | Within 48 hours after randomization
  Number of participants for whom corrective actions (e.g., potassium supplementation, fluid resuscitation) were implemented to allow safe administration of furosemide.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared. However, reasonable requests from qualified researchers will be considered after publication of the main results, subject to data use agreements and ethical approval

REFERENCES:
- [Derived] Beyls C, Mollet N, Gibert L, Huette P, Khamari M, Meynier J, Abou-Arab O, Mahjoub Y. Evaluation of natriuresis-guided depletion after cardiac surgery: protocol for a single-centre, open-label, randomised controlled trial-the EASY-CS study. BMJ Open. 2025 Oct 6;15(10):e108600. doi: 10.1136/bmjopen-2025-108600. PMID 41057198